CLINICAL TRIAL: NCT03761498
Title: Is There a Microbiome Associated With Poor Growth in Preterm Infants?
Status: Active, not recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Katherine Anne Stumpf, Assistant Professor of Pediatrics, University of Texas Southwestern Medical Center
Other Study IDs: STU 042018-061
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Growth Disorders; Growth Failure; Prematurity
MeSH Terms: conditions — Growth Disorders; Failure to Thrive; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Normal Growth: Require less than or equal to 110 kcal/kg/day to maintain growth curve
- Slow Growth: Require more than 110 kcal/kg/day to maintain growth curve
  Interventions: Other: Caloric Requirement

INTERVENTIONS:
Other: Caloric Requirement — Infants will be provided standard of care and given calories required to maintain appropriate growth per unit policies already in place.
  Groups: Slow Growth

SUMMARY:
This study evaluates the relationship between growth and stool microbiota in premature infants.

DETAILED DESCRIPTION:
Preterm infants often require increased caloric intake to maintain appropriate growth while in the neonatal intensive care unit (NICU). While some infants will have a clear source of need for greater calories, it is often not obvious why others require increased available calories to maintain appropriate growth. Emerging evidence suggests that patterns of gut microbiota may play a role in infant and childhood growth. We hypothesize that differences in the microbial pattern in preterm infants is related to poor growth and need for increased caloric intake. This may ultimately represent a therapeutic target to improve the growth of preterm infants in the NICU. This study aims to describe the differences in microbiome which may vary with growth pattern.

ELIGIBILITY:
Inclusion Criteria:

All infants less than 28 weeks gestation who are admitted to the Parkland Hospital NICU.

Exclusion Criteria:

Infants >27 weeks gestation. Infants with major congenital anomalies which may alter growth patterns.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Preterm infants born at less than 28 weeks gestation will be eligible from birth until discharge. Infants with major congenital anomalies which alter growth patterns will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
quantitative rT-PCR of stool microbiome | 8-10 weeks depending on length of stay in NICU
  alpha diversity of bacterial groups in normal growth vs. poor growth

CONTACTS AND LOCATIONS:
Locations (1):
- Parkland Hopsital and Health System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No